CLINICAL TRIAL: NCT03768167
Title: Posterolateral Corpectomy With Pyramesh Titanium Cage Reconstruction in Dorsolumber Metastatic Lesions
Brief Title: Corpectomy With Pyramesh Titanium Cage Reconstruction in Dorsolumber Metastatic Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, ahmed salaheldin mohammed saro, Assistant professor of neurosurgery, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sohag2
Record Dates: First submitted 2018-12-05; First posted 2018-12-07 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Spinal Metastases
Keywords: Corpectomy; Pyramesh; Posterolateral; Pediculectomy; Facetectomies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with metastatic spinal lesions (Other): corpectomy
  Interventions: Procedure: Posterolateral corpectomy

INTERVENTIONS:
Procedure: Posterolateral corpectomy — Investigators' goal in this study is to report clinical series of 26 patients in Sohag university hospital with dorsolumbar metastatic lesions from different primaries treated by single-stage posterolateral circumferential corpectomy with reconstruction by a pyramesh titanium cage and account the degree of improvement regarding the pain.

SUMMARY:
The vertebral column represents the most common bony site for metastasis with an incidence ranged from 30% to 70% in patients with metastatic neoplasms. The dorsal spine carries the highest frequent site for metastasis all over the vertebral column followed by the lumber spine. These metastatic lesions are clinical entities that often necessitate a complex spinal decompression and anterior reconstruction. Posterolateral approaches alone allow for excellent decompression with transpedicular fixation and safe visualization of the neural elements for corpectomy and reconstruction so the investigators can avoid the complications that can be happened with the staged surgery.

Purpose: investigators' aim in the study is to report cases and evaluate investigators' approach for fixation and assess the postoperative period regarding pain improvement and neurological deficit.

DETAILED DESCRIPTION:
At neurosurgery department in Sohag faculty of medicine, Between August 2014 and August 2017, 26 patients with single dorsolumbar metastatic spinal lesions with vertebral body collapse underwent a single-stage, circumferential corpectomy and anterior spinal reconstruction with a pyramesh titanium cage via a midline, posterior and lateral approach. Investigators included in the study patients with retropulsed fragment inside the canal that causes spinal cord compression with neurological manifestation. Metastatic work up was done for cases. Exclusion criteria include patients with more than one spinal metastases or extra-spinal metastasis, patients with other comorbidities as cardiac ill patients, patients with chronic renal failure and patients who received radiotherapy or chemotherapy within one year before surgery. A preoperative neurological assessment, full laboratory investigations were done. Investigators used the Quebec scale to assess the patients' improvement regarding pain, and muscle power scale to evaluate the motor.

ELIGIBILITY:
Inclusion Criteria:

* patients with retropulsed fragment inside the canal that causes spinal cord compression with neurological manifestation.

Exclusion Criteria:

* patients with more than one spinal metastases or extra-spinal metastasis.
* patients with other comorbidities as cardiac ill patients, patients with chronic renal failure.
* patients who received radiotherapy or chemotherapy within one year before surgery.

Ages: 33 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
(Quebec scale) to assess back pain in three years | 3 years
  (Quebec Scale) the lower scale the better is the pain
(muscle power grading scale) to evaluate motor power using in three years | 3 years
  (Muscle power grading) the higher the grade the better is the motor power

CONTACTS AND LOCATIONS:
Overall Officials: Roshdy A Elkhayat, Professor of neurosurgery, Study Chair — Assuit faculty of medicine
Locations (1):
- Ahmed Salaheldin Mohammed Saro, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No